CLINICAL TRIAL: NCT01092637
Title: School Age Outcomes Following a Newborn Cooling Trial
Brief Title: The TOBY Children Study
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: ISRCTN89547571; G0801320 (Other Grant/Funding Number: Medical Research Council (UK))
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Results first posted 2016-01-21 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2013-11

CONDITIONS: Cerebral Palsy; Hypoxia-Ischemia, Brain
MeSH Terms: conditions — Cerebral Palsy; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cooled: Child was allocated standard intensive care plus moderate whole body hypothermia treatment within 6 hours of birth
- Non-cooled: Child was allocated standard intensive care only within 6 hours of birth

SUMMARY:
The aim of this study is to determine the efficacy of therapeutic hypothermia following perinatal asphyxia on neurological and neuropsychological outcomes and also to assess academic attainment and any additional health, societal or educational costs associated with changes in outcome as a result of the intervention. This study will determine whether the apparent initial benefits of cooling are maintained in the longer term.

Perinatal asphyxia (a lack of oxygen occurring around the time of birth) may have long term consequences on brain functioning, which may be altered by treatment with hypothermia (cooling). Currently, there is no information on the effect of cooling on outcome beyond 18 months of age. We intend to assess at 6 - 7 years of age, the children that participated in the TOBY trial of whole body cooling following perinatal asphyxia and compare between the children that had received the cooling treatment soon after birth and those that were not treated with cooling, the number that survived with an intelligence quotient (IQ) greater than 84, the presence and severity of disabilities, educational attainment and the economic impact on families and service providers. If possible, children will be assessed in their school, with the option of alternative venues such as home or clinic if required.

During the assessment a paediatrician will conduct a neurological examination. A psychologist will administer psychometric tests to evaluate cognitive, behavioural and motor development. Questionnaires completed by parents and teachers will complete the data collection. Economic factors will also be assessed in the parent questionnaire.

Each child will have contact with the assessors during one school day with appropriate breaks. Assessments will take place over a period of 3 years.

DETAILED DESCRIPTION:
* Assessment tools used:

  * Wechsler Preschool and Primary Scale of Intelligence Third Edition (WPPSI-III; 2004) or Wechsler Intelligence Scales for Children
  * NEPSY Second Edition
  * Working Memory Test Battery for Children
* Neurological examination by paediatrician
* Questionnaire data from parents/guardians and teachers

ELIGIBILITY:
Inclusion Criteria:

* participant in the TOBY Study

Exclusion Criteria:

* previously documented instruction not to approach for inclusion in further TOBY projects

Ages: 72 Months to 87 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All participants were recruited to the TOBY randomised controlled trial as newborns, with confirmed moderate or severe hypoxic ischaemic encephalopathy.
  They were allocated either standard intensive care or standard intensive care plus moderate whole body hypothermia within 6 hours of birth.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2009-09; Primary Completion 2013-08 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Azzopardi, MD FRCPCH, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

REFERENCES:
- [Result] Azzopardi D, Strohm B, Marlow N, Brocklehurst P, Deierl A, Eddama O, Goodwin J, Halliday HL, Juszczak E, Kapellou O, Levene M, Linsell L, Omar O, Thoresen M, Tusor N, Whitelaw A, Edwards AD; TOBY Study Group. Effects of hypothermia for perinatal asphyxia on childhood outcomes. N Engl J Med. 2014 Jul 10;371(2):140-9. doi: 10.1056/NEJMoa1315788. PMID 25006720
- [Derived] Rivero-Arias O, Eddama O, Azzopardi D, Edwards AD, Strohm B, Campbell H. Hypothermia for perinatal asphyxia: trial-based resource use and costs at 6-7 years. Arch Dis Child Fetal Neonatal Ed. 2019 May;104(3):F285-F292. doi: 10.1136/archdischild-2017-314685. Epub 2018 Jul 11. PMID 29997167
- [Derived] Campbell H, Eddama O, Azzopardi D, Edwards AD, Strohm B, Rivero-Arias O. Hypothermia for perinatal asphyxia: trial-based quality of life at 6-7 years. Arch Dis Child. 2018 Jul;103(7):654-659. doi: 10.1136/archdischild-2017-313733. Epub 2018 Mar 6. PMID 29510998

RESULTS

PARTICIPANT FLOW:
Groups:
- Cooled: Child was allocated standard intensive care plus moderate whole body hypothermia treatment within 6 hours of birth. Cooling lasted for 72 hours then gradually rewarmed, after which normothermia was maintained.
  Between age 6 yr and 7 yr 3m child and family invited to participate in follow-up study.
  Questionnaire data collected from Parent(s) and Teacher(s). Paediatrician and Psychologist visited child in school or at home. Paediatrician neurodevelopmental examination completed and documented on Paediatrician Questionnaire.
  Psychologist completed the following tests:
  * Wechsler Pre-School and Primary Scale of Intelligence Third edition (WPPSI III)
  * NEPSY II selected sub-tests
  * Working Memory Test Battery for Children (WMTB-C)
  Assessors were blinded to original trial treatment allocation.
- Non-cooled: Child was allocated standard intensive care only within 6 hours of birth. Normothermia was maintained throughout.
  Between age 6 yr and 7 yr 3m child and family invited to participate in follow-up study.
  Questionnaire data collected from Parent(s) and Teacher(s). Paediatrician and Psychologist visited child in school or at home. Paediatrician neurodevelopmental examination completed and documented on Paediatrician Questionnaire.
  Psychologist completed the following tests:
  * Wechsler Pre-School and Primary Scale of Intelligence Third edition (WPPSI III)
  * NEPSY II selected sub-tests
  * Working Memory Test Battery for Children (WMTB-C)
  Assessors were blinded to original trial treatment allocation.
Period: Overall Study
Arm/Group | Cooled | Non-cooled
Started | 145 | 135
Completed | 98 | 86
Not Completed | 47 | 49
Not completed — Death | 47 | 49

BASELINE CHARACTERISTICS:
Population: 96 children died before school age assessment could take place. 184 children were included in the 6-7 year follow-up study, 98 cooled and 86 non-cooled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cooled | Non-cooled | Total
Number analyzed (Participants) | 145 | 135 | 280
Age, Continuous [Median (Full Range); unit: years] | 6.27 [6.03 to 8.82] | 6.24 [6.02 to 7.26] | 6.25 [6.02 to 8.82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 61 | 115
  Male | 91 | 74 | 165

OUTCOME MEASURES:

1. Primary Outcome: Number of Survivors With an IQ > 84
Description: IQ was measured using WPPSI III core tests
Time Frame: 7 years 3 months
Population: Children for whom IQ data at age 6-7 yr were available
Measure: Number; unit: participants
Groups:
- Cooled: Allocated cooling treatment at randomization to original trial. See full description in Participant flow section.
- Non-cooled: Allocated standard treatment (normothermia) at randomization to original trial. See full description in Participant flow section.
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 98 | 86
participants | 75 | 52

2. Secondary Outcome: Number of Survivors Without Disability
Description: IQ =>85, no neurological abnormalities, normal hearing, normal vision
Time Frame: 7 years 3 months
Population: Number of participants without disability. Two particpants in the cooled group and three in the non-cooled group could not be classified.
Measure: Number; unit: participants
Groups:
- Non-cooled: Allocated standard treatment (normothermia) at randomization. See full description in Participant flow section.
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 96 | 83
participants | 65 | 37

3. Secondary Outcome: Number of Survivors With Cerebral Palsy
Description: Number of participants diagnosed with Cerebral Palsy
Time Frame: 7 years 3 months
Population: Number of participants with cerebral palsy
Measure: Number; unit: participants
Arm/Group | Cooled | Non-cooled
Number analyzed (Participants) | 98 | 86
participants | 21 | 31

ADVERSE EVENTS:
Description: Serious and other adverse events were not collected/assessed
Arm/Group | Cooled | Non-cooled
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No